CLINICAL TRIAL: NCT01337427
Title: Optical Coherence Tomography (OCT) in a Multicenter, Randomized,Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate the Efficacy and Safety of PEGylated Interferon Beta-1a (BIIB017) in Subjects With Relapsing Multiple Sclerosis
Brief Title: Using Optical Coherence Tomography (OCT) to Evaluate the Efficacy and Safety of PEGylated Interferon Beta-1a (BIIB017) in Patients With Relapsing Multiple Sclerosis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was not feasible to conduct in the US and abroad.
Sponsor: Johns Hopkins University (Other)
Collaborators: Biogen (Industry)
Responsible Party: Peter Calabresi, MD, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00028117
Record Dates: First submitted 2011-04-07; First posted 2011-04-18 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: multiple sclerosis; relapsing; MS; injectable; subcutaneous; SC; PEGylated; interferon; PEG; OCT; Optical Coherence Tomography
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Placebo for 48 weeks, BIIB017 for 48 weeks (Placebo Comparator): Placebo every 2 weeks for 48 weeks followed by 125 mcg BIIB017 SC every 2 or 4 weeks for 48 weeks.
  Interventions: Drug: BIIB017
- BIIB017 every 2 weeks for 96 weeks (Experimental): 125 mcg BIIB017 SC every 2 weeks for 96 weeks.
  Interventions: Drug: BIIB017
- BIIB017 every 4 weeks for 96 weeks (Experimental): 125 mcg BIIB017 SC every 4 weeks for 96 weeks.
  Interventions: Drug: BIIB017

INTERVENTIONS:
Drug: BIIB017 — BIIB017 is supplied as a liquid in pre-filled syringes to deliver 0.5 mL of 0.25 mg/mL (125 mcg dose) of 20 kDa mPEG-O-2-methylpropionaldehyde-modified human IFN β-1a in 20 mM acetic acid/sodium acetate buffer pH 4.8, 150 mM arginine hydrochloride, and 0.005% Polysorbate 20.
  Other Names: PEGylated Interferon beta-1a; PEG IFN β-1a

SUMMARY:
This research sub-study is being completed as a part of the Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate the Efficacy and Safety of PEGylated Interferon Beta-1a (BIIB017) in Subjects with Relapsing Multiple Sclerosis (Protocol #: NA_00028117). This substudy is being done to understand the efficacy of BIIB017 by measuring the nerve fiber thickness in the eye.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
* A participant in the ADVANCE study aged 18 to 55 years old, inclusive, at the time of informed consent

Exclusion Criteria:

* As per the ADVANCE main study
* History of intraocular surgery, retinal disease, glaucoma, or diabetes
* Refractive errors of more than ±6.0 diopters
* Inability to tolerate OCT procedure

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
To determine the proportion of patients with RNFL decrease of 5 microns or more from baseline to month 12 in the BIIB-17 vs. placebo arms. | 1 year
To determine the proportion of patients with RNFL decrease of 5 microns or more from baseline to month 24 in the BIIB-17 vs. placebo arms. | 2 years

SECONDARY OUTCOMES:
Analysis of proportion of patients with a decrease of >10 percent of baseline value in any RNFL quadrant from baseline to month 12 in the BIIB-17 vs. placebo arms. | baseline and 1 year
Analysis of decrease between baseline scans and 3 month scan (to examine for pseudoatrophy) in this study population. | baseline and 3 months
Analysis of decrease between 3 month scans (mean and/or quadrant) and follow up scans (12 months) in this study population. | 3 months and 1 year
Analysis of macular volume decreases from baseline or 3 months to follow up scans at 12 months in this study population. | baseline and 1 year
Analysis of retinal nuclear layer decreases from baseline or 3 months to follow up scan at 12 months in this study population. | baseline and 1 year
Analysis of the above OCT parameters in patients with optic neuritis or history of optic neuritis. | 1 year
Analysis of proportion of patients with a decrease of >10 percent of baseline value in any RNFL quadrant from baseline to month 24 in the BIIB-17 vs. placebo arms. | baseline and 2 years
Analysis of decrease between 3 month scans (mean and/or quadrant) and follow up scans (24 months) in this study population. | 3 months and 2 years
Analysis of macular volume decreases from baseline or 3 months to follow up scans at 24 months in this study population. | baseline and 2 years
Analysis of retinal nuclear layer decreases from baseline or 3 months to follow up scan at 24 months in this study population. | baseline and 2 years
Analysis of the above OCT parameters in patients with optic neuritis or history of optic neuritis. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Calabresi, MD, Principal Investigator — Johns Hopkins University